CLINICAL TRIAL: NCT07353112
Title: Validation of the French Translation of SOSI-M in Healthy Children and in Children With Mild to Moderate Neurodevelopmental Disorder
Brief Title: Validation of the French Translation of the SOSI-M
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haute Ecole Ilya Prigogine (Other)
Responsible Party: Principal Investigator, Villa Lelia, Student, Haute Ecole Ilya Prigogine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUB2025977
Record Dates: First submitted 2025-12-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with neurodevelopmental disorders (NDD) (Experimental)
  Interventions: Diagnostic Test: Administration of the French translation of the SOSI-M test.
- Children with a neurotypical development (Experimental)
  Interventions: Diagnostic Test: Administration of the French translation of the SOSI-M test.

INTERVENTIONS:
Diagnostic Test: Administration of the French translation of the SOSI-M test. — Filmed administration of the French translation of the SOSI-M test
  We will then compare the scores of the two groups between them and with the scores obtained by other studies.
  There will be two operators that will evaluate each video 2 times (3 weeks between each evaluation) in order to mesure the metrologics qualities like fidelity.

SUMMARY:
The aim of this study is to validate the French version of the SOSI-M test on healthy children as well as on children with neurodevelopmental disorders (NDDs).

Therefore, the investigators will conduct a video recording of the test administration on a group of healthy children and on a group of children with NDDs.

The research question is: Is the French translation of the SOSI-M test equivalent, in terms of functionality and expected results, to the original version for a population of healthy children and children with mild to moderate neurodevelopmental disorders?

The hypothesis is that the psychometric properties of the French version are similar to those of the original version.

Secondly, the investigators will investigate: Does the difference in socio-cultural context between healthy Belgian and Senegalese children influence the SOSI-M score?

The hypothesis is that healthy Belgian children obtain better scores compared to healthy Senegalese children.

The scores of the two groups will be compared with each other and with those obtained in previous studies. Intra- and inter-rater reliability will also be assessed.

ELIGIBILITY:
For the groupe of children with neurodevelopmental disorders :

Inclusion criteria

* neurodevelopmental disorder (NDD)
* speak french and understand instructions in French
* and have not been assessed with the SOSI-M in the past 6 months.

Exclusion Criteria:

* Severe motor/cognitive impairment
* uncorrected visual/auditory impairment
* cerebral palsy diagnosis

For the neurotypical children :

Inclusion criteria :

- speak french and understand french instructions

Exclusion Criteria:

* diagnostic of musculoskeletal condition or neurodevelopmental or neurological condition
* health condition that contraindicates taking the SOSI-M

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
SOSI-M score | 1 day for the filmed passation of the french version of the sosi-m test.
  For the total raw score :
  0 = Abnormal 64 = Normal development of the child